CLINICAL TRIAL: NCT04127955
Title: Effectiveness of Theory of Planned Behavior Based Physical Activity Intervention Among 55-74 Years Turkish Adults Living in Nursing Home
Brief Title: A Nurse-led Theory of Planned Behavior Based Physical Activity Intervention Among Turkish Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Selma Baz, Instructor, Bahçeşehir University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IUC
Record Dates: First submitted 2019-10-08; First posted 2019-10-16 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2019-10

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Quasi-experimental design with one-group, pre-post test
  A nurse-led Theory of Planned Behavior based Physical Activity intervention consists of five component. These are a health education, a group walking, an individually tailored counseling session grounded on motivational interview technique, having the individuals keep track their physical activity levels with a pedometer, and use of physical activity pamphlet and posters as a reminder was planned. This intervention will be completed in eight weeks.
  Interventions: Other: Theory of Planned Behavior based Physical Activity Intervention

INTERVENTIONS:
Other: Theory of Planned Behavior based Physical Activity Intervention — Health education: The first component of intervention consisted of one session 30 minutes educational lesson relation to physical activity.
  Group walking: The format of the 15-minute group walking session included 5 minutes of warm-up, 5 minute moderate intensity walking, 5 minute cool-down.
  Counseling (individually tailored): The nurse received training about motivational interview technique for use in their physical activity counseling with participants. Using pedometers and step diary to set goals and monitor progress.
  Pedometer: pedometer will be used objective physical activity assessment. Measurement of physical activity levels, wearing a pedometer (Omron HJ321E) on a belt over one hip, all day for 7 days, removing for bathing and sleeping. A diary is also provided to record step count. The pedometer will be used for baseline and outcome measurement of step-counts for the trial.

SUMMARY:
The Theory of Planned Behavior has been successfully used in several programs to improve physical activity behavior. In this project, it is aimed to assess the effectiveness of Theory of Planned Behavior based physical activity intervention applied to 55-74 years old people living in nursing home in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study
* Aged 55 to 74
* Cognitive function of a score of greater than 24 on the Mini Mental State Examination
* Sedentary (Omaha system physical activity status ratings 1 or 2 score)
* To know Turkish literacy
* Time and go test score <14 seconds
* Approval of the resident's General Practitioner to participate

Exclusion Criteria:

* Uncontrolled cardiovascular, musculoskeletal or neurological disorders.
* Pain in motion or acute
* Communication barrier (due to hearing/vision impairment )
* > 3 falls in the previous year
* Need an walking aid (walkers, cane, crutches, walking sticks, etc.)

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in average daily steps | Average daily steps will be assessed intervention period at week 3-8 and 1 , 2 and 3 months follow-up visits.
  The number of steps weekly by the pedometer.
  The number of steps will be evaluated for the first time in the 3rd week of the intervention and each week until the end of the intervention (week 3-8).

SECONDARY OUTCOMES:
Changes in Blood Pressure | Blood pressure will be assessed baseline, before and after group walking and 1, 2 and 3 months follow-up visits
  Blood pressure will be assessed between baseline, before and after group walking and 1, 2, 3 months after the intervention using the upper arm blood pressure monitors (Omron M3 Comfort®, HEM-7134-E)
Changes in heart rate | Heart rate will be assessed baseline, before and after group walking and 1 , 2 and 3 months follow-up visits
  Heart rate will be assessed between baseline, before and after group walking and 1, 2, 3 months after the intervention using blood pressure monitors (Omron M3 Comfort®, HEM-7134-E)
Change in theory of planned behavior component | Baseline,3-month follow up.
  Theory of planned behavior components are including attitude, subjective norm, perceived behavior control, intention and behavior. The response used likert 1-7 format.
Change in The Problem Rating Scale | Change in physical activity will be assessed baseline, the week right after the intervention and 1 , 2 and 3 months follow-up visits
  The Omaha System include three components which are the Problem Classification Scheme, the Intervention Scheme, and the Problem Rating Scale for Outcomes. In this study, the Problem Rating Scale is used that evaluates the level of the problem and the results of the intervention. Change in physical activity measured with Omaha System Problem Rating Scale for Outcomes in which knowledge, behavior, status are rated on five-point Likert-type scales (1 = lowest / worse score, 5 = highest /best score). For example, a nurse may document a client's physical activity Knowledge as 1 (no knowledge), Behavior as 4 (Usually appropriate behavior), and Status as 2 (Severe signs/ symptoms).
Changes in health-related quality of life | Health-related quality of life will be assessed baseline, the week right after the intervention and 1, 2 and 3 months follow-up visits
  EQ-5D three-level version (EQ-5D-3L) descriptive systems is a five-dimensions questionnaire about the topics "mobility", "self-care", "usual-activities", "pain/discomfort" and "anxiety/depression".
Changes in EQ-VAS | Visual analogue scale (VAS) of EQ-5D Questionnaire will be assessed baseline, the week right after the intervention and 1, 2 and 3 months follow-up visits
  Visual analogue scale (VAS) of EQ-5D Questionnaire scaled from 0-100, corresponding to the worse and the best health imagined
Change in Body Mass Index (BKI) | BKI will be assessed baseline, the week right after the intervention and 3 months follow-up visit
  Weight (kg) will be measured using a balance scale with the measurement taken to the nearest 0.1 kg. Height (cm) will be measured using a stadiometer with the measurement taken to the nearest 0,5 cm. Weight and Height measurements will be then used to calculate the body mass index [BMI: Weight (kg) / (Height) 2 (m2)].
Change in waist hip ratio | Waist / hip ratio will be assessed baseline, the week right after the intervention and 3 months follow-up visit
  Waist circumference was measured at the level of the umbilicus to the nearest 0.1 cm. Hip circumference was measured at the level of the trochanter major. The waist / hip ratio was calculated as waist circumference (cm)/ hip circumference (cm).

CONTACTS AND LOCATIONS:
Overall Officials: Selda SEÇGİNLİ, PhD, Study Director — Istanbul University - Cerrahpasa